CLINICAL TRIAL: NCT02779582
Title: Oral Micronized Progesterone Effects on Perimenopausal Menstrual Flow: A Randomized, Double-masked, Placebo-controlled Trial
Brief Title: Oral Micronized Progesterone Effects on Perimenopausal Menstrual Flow
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jerilynn Prior, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H10-02975_1
Record Dates: First submitted 2015-12-10; First posted 2016-05-20 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Perimenopause; Menstrual Cramps
Keywords: Progesterone; Menstrual Flow
MeSH Terms: conditions — Dysmenorrhea | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone (Experimental): Oral micronized progesterone, 300 mg po daily, taken as three capsules daily before sleep for three months
  Interventions: Drug: Oral Micronized Progesterone
- Placebo (Placebo Comparator): Placebo, each taken as three capsules daily before sleep for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Micronized Progesterone — The dose of 300 mg of Progesterone is a physiological one that maintains the serum progesterone at or above the luteal (normal post-ovulatory) threshold for 24 hours. This duration of action is important because Progesterone is not safely taken during waking hours because of its soporific effects.
  Other Names: progesterone
  Arms: Progesterone
Drug: Placebo — pill with no effect
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the within-woman effect of oral micronized progesterone (Progesterone 300 mg at bedtime) on semi-quantitative menstrual flow measured by the DivaCup® (menstrual cup with volume indicators at 7.5, 15 and 30 ml) or by counting the number of soaked normal-sized sanitary products such as normal-sized tampons or pads as well as length of flow and frequency and severity of menstrual cramps (on a 0-4 scale) in women with hot flushes and night sweats who are qualified to enroll in the primary perimenopausal hot flush trial stratified by whether they are in Early or Late Perimenopause.

DETAILED DESCRIPTION:
The study will be a double-masked, placebo-controlled 28-day (4 week) baseline, 84-day (12 week) experimental trial, with a maximum number of 125 potential enrollees, with stratified random therapy assignment by Early or Late Perimenopause. Participants who meet the inclusion criteria for the original Progesterone for Perimenopausal Vasomotor Symptoms Study will be invited to join this additional sub-study. As part of the primary trial they will be randomly assigned into either the Progesterone or placebo group on a 1:1 basis. Primary and secondary data will be collected continuously throughout the study by completion of the Daily Perimenopause Diary-flow starting at baseline and continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* >35 to <58 years of age
* Willingness to participate in this sub-study
* Perimenopausal status either based on irregularity of menstrual periods, or by onset of hot flushes/night sweats in women with regular periods
* Ability and willingness to complete the -flow recording instrument
* Ability to understand, speak, read and write English.

Exclusion Criteria:

* Less than 35 or greater than 58 years of age
* More than 1-yr without menstrual flow at study enrollment, including those with a hysterectomy ± ovariectomy
* Peanut allergy (because peanut oil is used in the progesterone formulation)
* Current or recent (within 6-mo of study enrollment) use of hormonal therapies (estrogen, progesterone, progestin-releasing intrauterine device (IUD), hormonal contraceptives, hormonal fertility treatments), or plans to initiate use during the study period
* Planned pregnancy or fertility treatment during the study period
* Inability to understand, speak, read and write English

Ages: 35 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Amount of menstrual fluid | daily for four months

SECONDARY OUTCOMES:
Number of days of flow | daily for four months
Severity of menstrual cramps measured by a self-reported scale between zero and four (i.e. zero means 'no cramps' and four means 'very intense cramps') | daily for fourth months

CONTACTS AND LOCATIONS:
Overall Officials: Jerilynn C Prior, MD, FRCPC, Principal Investigator — UBC
Locations (1):
- Participation from home or in-person at University of British Columbia/Centre for Menstrual Cycle and Ovulation Research (CeMCOR)/Vancouver Coastal Health Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No